CLINICAL TRIAL: NCT01929603
Title: A Non-randomised, Open-label, Sequential, Multicentre, Two-part, Phase I Study to Assess the Effect of Rifampicin, a CYP Inducer, on the Pharmacokinetics of Olaparib Following Oral Dosing of a Tablet Formulation in Patients With Advanced Solid Tumours
Brief Title: Study to Assess the Effect of Rifampicin (CYP Inducer) on Blood Levels and Safety of Olaparib in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D0816C00008
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Solid Tumours
Keywords: oncology, cancer, tumour, anticancer drug, pharmacokinetics, olaparib, rifampicin, neoplasm, CYP P450 inducer
MeSH Terms: conditions — Neoplasms | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olaparib alone, olaparib+rifampicin (Experimental): Sequential treatments of olaparib alone followed by olaparib+rifampicin, with a washout period inbetween.
  Interventions: Procedure: Pharmacokinetic sampling; Drug: Rifampicin; Drug: Olaparib tablet dosing

INTERVENTIONS:
Procedure: Pharmacokinetic sampling — Blood sampling to measure olaparib, rifampicin and 4β-hydroxycholesterol
Drug: Rifampicin — Rifampicin (CYP inducer) 600mg taken once daily from Day 5 to Day 14 (Part A)
Drug: Olaparib tablet dosing — Olaparib 300mg tablet taken on Days 1 and 14 (Part A). Part B dosing is 300mg olaparib bi-daily

SUMMARY:
This is a 2-part study in patients with advanced solid tumours. Part A will investigate the effect of rifampicin on the PK parameters of olaparib in patients; Part B will allow patients continued access to olaparib after the PK phase and will provide additional safety data.

ELIGIBILITY:
Inclusion Criteria:-

For inclusion in the study, patients should fulfil the following criteria:

1. Provision of written informed consent prior to any study-specific procedures.
2. Patients aged greater than or equal to 18 years.
3. Histologically or, where appropriate, cytologically confirmed malignant solid tumour refractory or resistant to standard therapy or for which no suitable effective standard therapy exists.

4 Patients must have normal organ and bone marrow function measured within 28 days prior to administration of investigational product (IP) as defined below: Haemoglobin (Hb) greater than or equal to 10.0 g/dL, with no blood transfusions in the previous 28 days.

Absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L. White blood cells (WBC) greater than 3 x 109/L. Platelet count greater than or equal to 100 x 109/L. Total bilirubin less than or equal to 1.5 x institutional upper limit of normal (ULN) (except in the case of Gilbert's disease).

Aspartate aminotransferase (AST), alanine aminotransferase (ALT) less than or equal to 2.5 x institutional ULN unless liver metastases are present, in which case it must be less than or equal to 5x ULN, Serum creatinine less than or equal to 1.5 x institutional ULN.

5. Calculated serum creatinine clearance greater than 50 mL/min (using Cockroft-Gault formula or by 24 hour urine collection).

6. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.

7. Patients must have a life expectancy of greater than or equal to 16 weeks. 8. Evidence of non-childbearing status for women of childbearing potential, or post menopausal status: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on Day 1 of Part A. Post-menopausal is defined as: Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments.

Luteinising hormone and follicle stimulating hormone levels in the post menopausal range for women under 50 years of age.

Radiation-induced oophorectomy with last menses greater than 1 year ago. Chemotherapy-induced menopause with greater than 1 year interval since last menses.

Surgical sterilisation (bilateral oophorectomy or hysterectomy). 9. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

10. Patients must be on a stable concomitant medication regimen (with the exception of electrolyte supplements), defined as no changes in medication or in dose within the 2 weeks prior to start of olaparib dosing, except for bisphosphonates, denosumab, and corticosteroids, which should be at a stable dose for at least 4 weeks prior to the start of olaparib dosing.

Exclusion Criteria:- Patients should not enter the study if any of the following exclusion criteria are fulfilled.

1. Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff, its agents, and/or staff at the study site).
2. Previous enrolment in the present study.
3. Participation in another clinical study with an IP during the last 14 days (or a longer period depending on the defined characteristics of the agents used).
4. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 2 weeks prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study, as long as these were started at least 4 weeks prior to treatment.
5. Patients who have received or are receiving inhibitors or inducers of CYP3A4.
6. Toxicities (greater than or equal to Common Toxicity Criteria for Adverse Events [CTCAE] Grade 2) caused by previous cancer therapy, excluding alopecia.
7. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of the IP until the end of Part A.
8. Patients with brain metastases. A scan to confirm the absence of brain metastases is not required.
9. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of major surgery.
10. Patients considered a poor medical risk due to a serious uncontrolled medical disorder, non malignant systemic disease, uncontrolled seizures, or active uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive bilateral interstitial lung disease on high resolution computer tomography (HRCT) scan, or any psychiatric disorder that prohibits obtaining informed consent.
11. Patients who have diabetes mellitus.
12. Patients who have gastric, gastro-oesophageal, or oesophageal cancer .
13. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders or significant gastrointestinal resection likely to interfere with the absorption of olaparib.
14. Breastfeeding women.
15. Immunocompromised patients, eg, patients who are known to be serologically positive for human immunodeficiency virus (HIV).
16. Patients with known active hepatic disease (eg, hepatitis B or C).
17. Patients with a known hypersensitivity to rifampicin or any of the excipients of the product.
18. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
19. Resting electrocardiogram (ECG) at screening with measurable QT interval (QT) corrected for heart rate (QTc) greater than 470 msec at 2 or more time points within a 24 hour period or family history of long QT syndrome.
20. Concomitant medication contraindicated for use with rifampicin (including, but not limited to): atazanavir, darunavir, fosamprenavir, ritonavir-boosted saquinavir, saquinavir, or tipranavir.
21. Patients who have jaundice.
22. Patients who weigh less than 50 kg.
23. Clinical judgment by the investigator that the patient should not participate in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of olaparib by assessment of maximum plasma olaparib concentration (Cmax) | Blood samples are collected on olaparib dosing days (Day 1 and 14) at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A.
  Rate and extent of absorption of olaparib following single oral doses of olaparib tablet formulation by assessment of maximum plasma olaparib concentration (Cmax). Olaparib doses are first without, then with rifampicin.
Pharmacokinetics of olaparib by assessment of area under the plasma concentration time curve from zero to infinity (AUC) | Blood samples are collected on olaparib dosing days (Day 1 and 14) at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A.
  Rate and extent of absorption of olaparib following single oral doses of olaparib tablet formulation by assessment of area under the plasma concentration time curve from zero to infinity (AUC).
  Olaparib doses are first without, then with rifampicin.
Pharmacokinetics of olaparib by assessment of area under the plasma concentration time curve from zero to the last measurable time point, AUC0-t, if AUC is not adequately estimable. | Blood samples are collected on olaparib dosing days (Day 1 and 14) at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A.
  Rate and extent of absorption of olaparib following single oral doses of olaparib tablet formulation by assessment of area under the plasma concentration time curve from zero to the last measurable time point, AUC0-t, if AUC is not adequately estimable. Olaparib doses are first without, then with rifampicin.

SECONDARY OUTCOMES:
Pharmacokinetics of olaparib by assessment of time to reach maximum plasma concentration for olaparib (tmax). | Blood samples are collected on olaparib dosing days (Day 1 and 14) at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A.
  Rate and extent of absorption of olaparib following single oral doses of olaparib tablet formulation by assessment of time to reach maximum plasma concentration for olaparib (tmax). Olaparib doses are first without, then with rifampicin.
Pharmacokinetics of olaparib by assessment of olaparib area under the plasma concentration time curve from zero to the last measurable time point (AUC0-τ). | Blood samples are collected on olaparib dosing days (Day 1 and 14) at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A.
  Rate and extent of absorption of olaparib following single oral doses of olaparib tablet formulation by assessment of olaparib area under the plasma concentration time curve from zero to the last measurable time point (AUC0-τ). Olaparib doses are first without, then with rifampicin.
Pharmacokinetics of olaparib by assessment of olaparib apparent clearance (CL/F). | Blood samples are collected on olaparib dosing days (Day 1 and 14) at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A.
  Rate and extent of absorption of olaparib following single oral doses of olaparib tablet formulation by assessment of olaparib apparent clearance (CL/F). Olaparib doses are first without, then with rifampicin.
Pharmacokinetics of olaparib by assessment of olaparib apparent volume of distribution (Vz/F). | Blood samples are collected on olaparib dosing days (Day 1 and 14) at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A.
  Rate and extent of absorption of olaparib following single oral doses of olaparib tablet formulation by assessment of olaparib apparent volume of distribution (Vz/F). Olaparib doses are first without, then with rifampicin.
Pharmacokinetics of olaparib by assessment of olaparib terminal half-life (t1/2). | Blood samples are collected on olaparib dosing days (Day 1 and 14) at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A.
  Rate and extent of absorption of olaparib following single oral doses of olaparib tablet formulation by assessment of olaparib terminal half-life (t1/2). Olaparib doses are first without, then with rifampicin.
Pharmacokinetics of rifampicin by assessment of plasma concentrations of rifampicin during rifampicin dosing period. | Rifampicin is dosed daily from Days 5 to 17 in Part A. Blood samples are collected on Days 5, 9, 14 and 17 at 2 hours post rifampicin dose
  Rate and extent of absorption of rifampicin following multiple doses of rifampicin by assessment of plasma concentrations of rifampicin during rifampicin dosing period.
Demonstration of induction of CYP by assessment of plasma concentrations of 4β-hydroxycholesterol during rifampicin dosing period. | Blood samples are collected on Days 5, 9, 14 and 17 at pre-dose of rifampicin in Part A
  Demonstration of CYP induction by assessment of plasma concentrations of 4β-hydroxycholesterol during rifampicin dosing period.
Assessment of the safety and tolerability of olaparib by collection of adverse event reports | Part A: From baseline, every visit until 30 days after last dose. Part B, from start to 12 months after the last patient has entered Part B
  Assessment of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Determine safety and tolerability of olaparib by assessment of 12 lead electrocardiograms | Part A: baseline, Days -1, 17 (and within 30 days post last olaparib dose if not in Part B).
  Assessment of standard 12 lead electrocardiograms (ECGs)
Determine safety and tolerability of olaparib by physical examination | Part A: baseline, Day -1 and within 30 days after last dose. Part B: Day 1.
  Assessment of physical examination
Determine safety and tolerability of olaparib by assessment of vital signs | Part A: baseline, Days 1,2 and 3. Part B: Days 1,8,15,22,29 then every 4 weeks. Final assessment within 30 days after last dose.
  Assessment of standard vital signs (including blood pressure, pulse)
Determine safety and tolerability of olaparib by assessment of clinical chemistry results | Part A: baseline, Days -1, 9, 14, 17. Part B: Days 1,8,15,22,29 then every 4 weeks. Final assessment within 30 days after last dose.
  Assessment of laboratory parameters (clinical chemistry)
Determine safety and tolerability of olaparib by assessment of haematology results | Part A: baseline, Days -1, 9, 14, 17. Part B: Days 1,8,15,22,29 then every 4 weeks. Final assessment within 30 days after last dose.
  Assessment of laboratory parameters (haematology)
Determine safety and tolerability of olaparib by assessment of urinalysis results | Part A: baseline, Days -1, 14, 17. Part B: Day 1 only
  Assessment of laboratory parameters (urinalysis)

CONTACTS AND LOCATIONS:
Overall Officials: Anitra Fielding, Study Director — AstraZeneca Senior Research Physician; Luc Dirix, Principal Investigator — GZA Ziekenhuizen Campus Sint-Augustinus
Locations (5):
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Wilrijk
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht

REFERENCES:
- [Derived] Dirix L, Swaisland H, Verheul HM, Rottey S, Leunen K, Jerusalem G, Rolfo C, Nielsen D, Molife LR, Kristeleit R, Vos-Geelen J, Mau-Sorensen M, Soetekouw P, van Herpen C, Fielding A, So K, Bannister W, Plummer R. Effect of Itraconazole and Rifampin on the Pharmacokinetics of Olaparib in Patients With Advanced Solid Tumors: Results of Two Phase I Open-label Studies. Clin Ther. 2016 Oct;38(10):2286-2299. doi: 10.1016/j.clinthera.2016.08.010. Epub 2016 Oct 10. PMID 27745744
- See also: D0816C00008_Study_Synopsis_Redacted.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1867&filename=D0816C00008_Study_Synopsis_Redacted.pdf